CLINICAL TRIAL: NCT04327427
Title: Outcome Analysis of Antiplatelet Therapy With Aspirin in Liver Transplantation
Brief Title: Outcome Analysis of Aspirin in Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01889
Record Dates: First submitted 2020-03-17; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Liver Transplant; Complications
Keywords: liver transplantation; aspirin; tumor recurrence; HCC; graft survival
MeSH Terms: conditions — Recurrence | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Aspirin — Outcome Analysis of Aspirin in liver transplantation

SUMMARY:
In the experimental setting inhibition of platelet activation was able to reduce immune-mediated necroinflammatory liver disease and consecutively hepatocellular carcinoma development. Therefore, antiplatelet therapy may not only have a preventive effect on hepatic artery patency but also on tumor recurrence.

So far and to the best of our knowledge, no study investigated the effect of antiplatelet therapy on hepatic arterial patency, tumor recurrence and graft survival after primary liver transplantation.

DETAILED DESCRIPTION:
Outcome Analysis of antiplatelet therapy with Aspirin in Liver Transplantation

BACKGROUND Arterial complications after liver transplantation (LT) are still one of the most serious complications, which might result in liver necrosis, abscess formation, ischemic cholangiopathy, and eventually graft loss. The sequel of these adverse events has a negative impact on graft and patient survival and remains a life-threatening complication with a high mortality and retransplantation rate. Therefore, an uncompromised inflow of the hepatic artery is crucial to avoid any occlusion after LT.

In the literature, the incidence of hepatic artery thrombosis ranges between 2.5 and 10%. So far, the possibility of preventing hepatic artery thrombosis through specific pharmacological prophylaxis with antiplatelet agents (Aspirin) has been poorly investigated, which may be in part due to the impaired coagulative state at the time of transplantation and the early postoperative period. On the other hand, platelets, the chief effectors of vascular homeostasis, have been identified as important players in the pathogenesis of both acute and chronic liver diseases in animal models.

In the experimental setting inhibition of platelet activation was able to reduce immune-mediated necro-inflammatory liver disease and consecutively hepatocellular carcinoma development. Therefore, antiplatelet therapy may not only have a preventive effect on hepatic artery patency but also on tumor recurrence.

So far and to the best of our knowledge, no study investigated the effect of antiplatelet therapy on hepatic arterial patency, tumor recurrence and graft survival after primary liver transplantation.

STUDY OBJECTIVES The primary goal of this study is to conduct a multicentre cohort analysis to investigate whether antiplatelet therapy with Aspirin has an impact on hepatic arterial patency after primary liver transplantation.

Specific aim #1: To evaluate if antiplatelet therapy with Aspirin has a protective effect on arterial patency after primary LT.

Specific aim #2: To identify if antiplatelet therapy with Aspirin has a protective effect on acute cellular rejection.

Specific aim #3: To identify if antiplatelet therapy with Aspirin has protective effect on tumor recurrence (HCC).

Specific aim #4: To investigate whether antiplatelet therapy with Aspirin has a protective effect on graft survival.

STUDY DESIGN This will be a multicentre single cohort study including only cases of deceased donor primary liver transplantation. Primary endpoint is 30-day arterial patency in patients with or without antiplatelet therapy with Aspirin after liver transplantation. Secondary endpoints include postoperative complications, tumor recurrence, graft- and patient survival. The study protocol has received approval by the local ethics committee (2016-01889) as well as published here prior to data collection.

SETTING This multicentre cohort study will include several high-volume centres worldwide. Each participating centre requires a prospective database from that data can be extracted. All consecutive cases of deceased donor liver transplantation requiring from 1st of January 2013 until 31st of December 2015 are included allowing a minimum follow-up time of 24 months. Data collection at Aspirin4olt.org will be prospective, structured, anonymized, and encrypted.

PUBLICATION POLICY For upcoming publications, two authorships of the participating centres will be guaranteed as a group-authorship indexed in PubMed.

INSTITUTIONAL REVIEW POLICY / ETHICAL POLICY Each participating centre is responsible to contact their local ethics committee and receive approval for participation, if applicable. For example, this project is considered as an audit in some countries and thus there is no need for formal approval in the form of a protocol submission.

ELIGIBILITY CRITERIA

Inclusion criteria:

Adult Liver transplantation (age ≥18 years) Deceased donor after brain death (DBD) or deceased donor after circulatory death (DCD) Primary liver transplantation, whole graft Arterial anastomosis: end-to-end, back table reconstruction

Exclusion criteria:

Split liver and living donor liver transplantation Paediatric liver transplantation (recipient age <18 years) Arterial conduits Multivisceral transplantations Retransplantations

ESTIMATED SAMPLE SIZE Each centre should provide at least 30 cases that meet the inclusion criteria to allow adequate event rates for each outcome.

Statistical methods The primary and secondary endpoints will be compared with patient and operation characteristics with univariate analysis. ROC Curve analysis will be performed to dichotomize continuous variables. Multivariable analysis (binary logistic and Cox regression) will be performed to identify independent risk factors. Statistical analysis will be performed using R Studio version 1.0.44 (RStudio, Inc. GNU Affero General Public License v3, Boston, MA, 2016) with the graphical user interface rBiostatistics.com beta version (rBiostatistics.com, London, UK, 2017, GNU License).

Christian E. Oberkofler Philip C. Müller Dimitri A. Raptis Henrik Petrowsky On behalf of the Aspirin4olt.org team Swiss HPB Center, Department of Surgery and Transplantation, University Hospital Zurich, Switzerland

ELIGIBILITY:
Inclusion Criteria:

* Adult Liver transplantation(age ≥18 years)
* Deceased donor after brain death (DBD) or deceased donor after circulatory death (DCD)
* Primary liver transplantation, whole graft
* Arterial anastomosis: end-to-end, back table reconstruction

Exclusion Criteria:

* Split liver and living donor liver transplantation
* Paediatric liver transplantation (recipient age <18 years)
* Arterial conduits
* Multivisceral transplantations
* Retransplantations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicentrecohort study will include several high-volume centresworldwide. Each participating centrerequires a prospective database from that data can be extracted. All consecutive cases of deceased donor liver transplantation requiring from 1stofJanuary 2013until 31stof December 2015are included allowing a minimum follow-up time of 24months.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Aspirin and arterial patency | 2 years
  We will look, if antiplatelet therapy with Aspirin has a protective effect on arterial patency after primary liver transplantation by looking at postoperative lab values and imaging, if they were perfromed.

SECONDARY OUTCOMES:
Aspirin and cellular rejection | 2 years
  We will analyze patients with and without postoperative cellular rejection and the intake of Aspirin.
Aspirin and tumor recurrence | 2 years
  We will look at post transplant tumor recurrence and if the recurrence does correlate with Aspirin intake.
Aspirin and graft survival | 2 years
  We will look at the postoperative graft survival and devide graft survival in the group of patients who were under Aspirin postoperative with those who did not take Aspirin postoperative; both groups will be then compared.

CONTACTS AND LOCATIONS:
Overall Officials: Christian E Oberkofler, MD, Principal Investigator — University of Zurich
Locations (1):
- Department of Visceral and Transplantation Surgery, Zurich, CH/Zürich, Switzerland

IPD SHARING:
Plan to Share IPD: No